CLINICAL TRIAL: NCT01313793
Title: A Phase 1 Open-Label Study Of Pf-00299804 In Healthy Volunteers To Demonstrate The Bioequivalence Of The Proposed Commercializable Formulation Administered As One 45-Mg Tablet Relative To Three 15-Mg Clinical Formulation Tablets
Brief Title: A Bioequivalence (BE) Study Comparing The Commericializable And Clinical Formulations Of PF-00299804
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A7471022
Record Dates: First submitted 2011-02-08; First posted 2011-03-14 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence (BE) Study; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects will receive clinical formulation (treatment A) followed by commercializable formulation (treatment B).
  Interventions: Drug: Treatment A-B
- Sequence 2 (Experimental): Subjects will receive commercializable formulation (treatment B) followed by clinical formulation (treatment A).
  Interventions: Drug: Treatment B-A

INTERVENTIONS:
Drug: Treatment A-B — Subjects to receive 3 X 15 mg tablets of the clinical formulation in first period then 1 x 45 mg tablet of the commericializable formulation in 2nd period.
  Arms: Sequence 1
Drug: Treatment B-A — Subjects to receive 1 x 45 mg tablet of the commericializable formulation in first period then 3X 15 mg tablets of the clinical formulation in 2nd period.
  Arms: Sequence 2

SUMMARY:
The study will determine if bioequivalence can be claimed between the proposed commericializable formulation and the current clinical formulation. Specifically, if the 90% confidence intervals of the ratio for Area under the curve (AUC) and maximum concentration (CMax) are within the 80%-125% guidance limits.

DETAILED DESCRIPTION:
A bioequivalence (BE) study between two formulations of PF-00299804.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects including males between the ages of 18 and 55 years and/or females of non childbearing potential between the ages of 18 and 55 years. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant dermatologic, hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* Use of tobacco- or nicotine- containing products (or a positive urine drug cotinine test).
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication.
* 12 lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Pregnant or nursing females and females of childbearing potential including those with tubal ligation. To be considered for enrollment, women of 45 to 55 years of age who are postmenopausal (defined as being amenorrheic for at least 2 years) must have confirmatory FSH test results at Screening.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication. Depo Provera must be discontinued at least 6 months prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of less than 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf of of PF 00299804 | 6-8 weeks
AUClast of PF 00299804 | 6-8 weeks
Cmax of PF 00299804 | 6-8 weeks

SECONDARY OUTCOMES:
Plasma AUCinf of PF 00299804. | 6-8 weeks
CL/F of PF 00299804. | 6-8 weeks
Tmax of PF 00299804. | 6-8 weeks
tlast of PF 00299804. | 6-8 weeks
t1/2 of PF 00299804. | 6-8 weeks
Plasma AUCinf of PF-05199265 | 6-8 weeks
AUClast of PF-05199265 | 6-8 weeks
Cmax of PF-05199265 | 6-8 weeks
Tmax of PF-05199265 | 6-8 weeks
tlast of PF-05199265 | 6-8 weeks
Safety laboratory tests, physical examination, concomitant medication and adverse event monitoring | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471022&StudyName=A%20Bioequivalence%20%28BE%29%20Study%20Comparing%20The%20Commericializable%20And%20Clinical%20Formulations%20Of%20PF-00299804